CLINICAL TRIAL: NCT02497248
Title: PERSONALIZE-AF: Non-invasive Characterization of the Mechanisms of Atrial Fibrillation
Brief Title: Non-invasive Characterization of the Mechanisms of Atrial Fibrillation Maintenance
Acronym: PERSONALIZE
Status: Completed | Type: Observational
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Collaborators: Universitat Politècnica de València (Other); Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Other Study IDs: PERSONALIZE-AF
Record Dates: First submitted 2015-06-30; First posted 2015-07-14 (Estimated); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Pulmonary Vein Ablation; Mitral stenosis; Body surface mapping
MeSH Terms: conditions — Atrial Fibrillation; Mitral Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- - Patients with paroxysmal AF.: Patients with AF episodes that terminates spontaneously or with intervention in less than seven days with clinical indication of pulmonary vein ablation.
  Interventions: Procedure: Pulmonary vein ablation
- - Patients with persistent AF.: Patients with AF episodes that fails to self-terminate within seven days or require pharmacologic or electrical cardioversion to restore sinus rhythm with clinical indication of pulmonary vein ablation..
  Interventions: Procedure: Pulmonary vein ablation
- - Patients with mitral stenosis.: - Patients with mitral stenosis and clinical indication for AF ablation undergoing percutaneous balloon mitral valvuloplasty (PBMV) with clinical indication of pulmonary vein ablation..
  Interventions: Procedure: Pulmonary vein ablation

INTERVENTIONS:
Procedure: Pulmonary vein ablation — Simultaneous biatrial endocardial electroanatomical mapping by high-density basket catheter (64 pin) and customized body surface mapping (57 electrodes) followed by circumferential pulmonary vein ablation.
  Other Names: Mitral Valvuloplasty in patients with severe mitral stenosis

SUMMARY:
Currently available antiarrhythmic drugs for the treatment of atrial fibrillation (AF) have a limited efficacy and often cause long-term side effects. Pulmonary vein isolation is the therapy of choice in drug-refractory patients. Recent studies have shown that ablation have a greater efficacy in patients in whom AF is maintained hierarchically and after ablation of rotors. The non-invasive identification of specific mechanism of AF maintenance in each patient could allow the selection of the most appropriate treatment.

DETAILED DESCRIPTION:
The MAIN GOAL of this project is to clinically validate the technology for the noninvasive identification of the mechanisms responsible for maintenance of AF by body surface electrical mapping. To achieve this goal, noninvasive mapping of the atrial activity will be correlated with simultaneous endocardial mapping (high density contact catheters) using advanced signal analyses techniques (Dominant frequency, phase and causality mapping, inverse solution problem). These analyses will be performed in patients with different mechanisms of maintenance of AF (e.g. paroxysmal, persistent, valvular) undergoing AF ablation for clinical indication. Both endocardial and body surface mapping results will be correlated with biomarkers levels, MRI scans and AF outcomes of AF ablation at 6 months and 1 year after the procedure.

Wide antrum circumferential pulmonary vein isolation with demonstration of bidirectional block will be performed using standard cooled-tip radiofrequency catheters. In patients with mitral stenosis, PBMV will be performed according to Inoue´s technique followed by wide antrum circumferential pulmonary vein isolation. In all patients, MRI/CT scans and fibrosis biomarkers will be obtained at baseline, 6 months and 1 year post ablation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with paroxysmal AF symptomatic and refractory to at least one antiarrhythmic medication.
* Patients with persistent AF symptomatic and refractory to at least one antiarrhythmic medication.
* Patients with severe mitral stenosis (mitral valve area ≤1.5 cm2, stage D) and favorable valve morphology in the absence of left atrial thrombus or moderate-to-severe mitral regurgitation.
* Patients must be able and willing to provide written informed consent to participate in the study.
* Prior anticoagulation for> 4 weeks or transesophageal echocardiogram excluding intracardiac thrombi (in patients with paroxysmal AF).

Exclusion Criteria:

* Patients with inadequate anticoagulation levels.
* Patients with left atrial thrombus, tumor, or another abnormality which precludes catheter introduction on TEE prior to the procedure.
* Patients with moderate-to-severe mitral regurgitation.
* Patients with contraindications to systemic anticoagulation with heparin or coumadin.
* Prior atrial fibrillation ablation.
* Patients who are or may potentially be pregnant.
* Contraindication for adenosine administration;
* Current enrollment in another investigational drug or device study.
* Pacemaker or Implantable Cardioverter Defibrillator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AF patients with different mechanisms of maintenance (i.e. paroxysmal, persistent, valvular) and clinical indication for AF ablation.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Freedom from atrial fibrillation off antiarrhythmic medications in patients with either paroxysmal, persistent AF or valvular stenosis AF. | 12 months post-first ablation procedure

SECONDARY OUTCOMES:
Freedom from atrial fibrillation on or off antiarrhythmic medication post-first ablation procedure and after redo procedures. | at 6 and 12 months
Freedom from atrial fibrillation and other atrial arrhythmias post-first ablation procedure and after redo procedures. | at 6 and 12 months
Incidence of peri-procedural complications | during ablation procedure and 12 months after
Procedure duration | Duration of ablation procedure, and valvuloplasty if indicated, in minutes
Body surface recording analysis by 120 disposable electrodes distributed over the patient's chest and connected to the polygraph. | During ablation procedure, and valvuloplasty if indicated
Electroanatomic reconstruction and recordings of electrical activity: a three-dimensional reconstruction of atrium and coronary sinus is obtained using high density catheters and an electroanatomic navigation system. | During ablation procedure, and valvuloplasty if indicated
Atrial fibrosis determination using late gadolinium enhancement-MRI | At 6 and 12 months
Fluoroscopy time | During ablation procedure, and valvuloplasty if indicated, in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Atienza, MD, Principal Investigator — Red de Investigación Cardiovascular
Locations (1):
- Felipe Atienza Fernandez, Madrid, Spain

REFERENCES:
- [Background] Atienza F, Almendral J, Ormaetxe JM, Moya A, Martinez-Alday JD, Hernandez-Madrid A, Castellanos E, Arribas F, Arias MA, Tercedor L, Peinado R, Arcocha MF, Ortiz M, Martinez-Alzamora N, Arenal A, Fernandez-Aviles F, Jalife J; RADAR-AF Investigators. Comparison of radiofrequency catheter ablation of drivers and circumferential pulmonary vein isolation in atrial fibrillation: a noninferiority randomized multicenter RADAR-AF trial. J Am Coll Cardiol. 2014 Dec 16;64(23):2455-67. doi: 10.1016/j.jacc.2014.09.053. PMID 25500229